CLINICAL TRIAL: NCT07053020
Title: A Phase 1b/2 Open-label, Dose-ranging Safety and Efficacy Study of Oral Cladribine in Patients With Acute Myeloid Leukemia (AML)
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-1896; NCI-2025-04733 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2025-06-30; First posted 2025-07-08 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-06

CONDITIONS: Acute Myeloid Leukemia (AML)
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Cytarabine; Cladribine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Part 1/2 Treatment with Oral Cladribine in Patients with Acute Myeloid Leukemia (Experimental): Participants may be in the hospital up to the first 5 days on study to all monitoring for tumor lysis syndrome (TLS) and toxicities.
  Interventions: Drug: Cytarabine; Drug: Oral Cladribine

INTERVENTIONS:
Drug: Cytarabine — Given by intravenous adminstration
Drug: Oral Cladribine — Given Orally

SUMMARY:
The goal of Part 1 of this clinical research study is to find the highest tolerable dose of cladribine that can be given in combination with low dose cytarabine (LDAC) and venetoclax to patients who have AML.

The goal of Part 2 of this clinical research study is to learn if the dose of cladribine found in Part 1, when combined with LDAC and venetoclax, can help to control the disease.

DETAILED DESCRIPTION:
Primary Objective:

The primary objective of Phase 1 is to determine safety and tolerability of oral cladribine in patients with AML and to identify a RP2D.

Secondary Objective:

The secondary objectives of Phase 1 are to provide a qualitative assessment of systemic exposure based on plasma cladribine concentrations after administration of oral cladribine to patients with AML and to explore the activity of cladribine/LDAC/venetoclax in patients with relapsed or refractory AML.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of written informed consent prior to any study related procedures.
2. Disease characteristics, defined as:

   Part 1:

   Dose-escalation cohorts: Patients with relapsed and/or refractory AML.

   Part 2:

   Cohort A: Patients aged .18 years with newly diagnosed ts-AML, defined as patients with prior diagnosis of MDS, treated with hypomethylating agents who have then progressed to AML. Prior therapy with hydroxyurea, hematopoietic growth factors, HMA, ATRA, or a total dose of cytarabine up to 2g (for emergency use for stabilization) is allowed.

   Cohort B: Patients aged . 60 years with newly diagnosed AML with monocytic phenotype, defined as AML-M5 by FAB or flow cytometry, and/or patients . 60 years with newly diagnosed AML with RAS mutations. Patients aged < 60 years who are unsuitable for standard induction therapy may be eligible after discussion with primary investigator.
3. Adequate renal and hepatic organ function as indicated by the following laboratory values:

   * Serum creatinine . 2.0xupper limit of normal (ULN)
   * Serum total bilirubin .2xULN (with the exception of patients with known Gilbert's syndrome: serum total bilirubin must be <3xULN in these patients)
   * Aspartate aminotransferase (serum glutamic oxaloacetic transaminase) and alanine aminotransferase (serum glutamic pyruvic transaminase) .2.5xULN or .5xULN if due to leukemic involvement)
4. Adequate cardiac function with a left ventricular ejection fraction .50%
5. Female participants are eligible to enter and participate in the study if they are of nonchildbearing potential. Female participants of childbearing age must use at least 2 forms of effective birth control during the study treatment period and for at least 90 days after the last dose of investigational product.
6. Male participants are eligible to enter and participate in the study if they agree to use effective methods of contraception during the study treatment period and for at least 90 days after the last dose of investigational product.

Exclusion Criteria:

1. Uncontrolled intercurrent illness including, but not limited to ongoing or active uncontrolled infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
2. History of allergic reactions attributed to compounds of similar chemical or biologic composition to any of the compounds in the study.
3. Legal incapacity or limited legal capacity.
4. Inability to swallow oral medications (capsules and tablets) without chewing, breaking, crushing, opening or otherwise altering the product formulation.
5. Patients unwilling to comply with protocol requirements related to the assigned part.
6. Patients with psychiatric illness/social situations that would limit compliance with study requirements.
7. Pregnant women are excluded from this study because the agents used in this study have the potential for teratogenic or abortifacient effects. Because there is a potential risk for adverse events in nursing infants secondary to treatment of the mother with chemotherapy agents, breastfeeding should also be avoided.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2028-06-30 (Estimated); Study Completion 2030-06-30 (Estimated)

PRIMARY OUTCOMES:
Safety and Adverse Events (AEs) | Through study completion; an average of 1 year
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Gautam Borthakur, MBBS, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- The University of Texas M. D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org